CLINICAL TRIAL: NCT02602496
Title: Promoting Gastrointestinal Health and Reducing Subclinical Inflammation in Obese Individuals Through Intake of Whole Wheat Products in Comparison With Fruits and Vegetables
Brief Title: Promoting Gastrointestinal Health and Reducing Subclinical Inflammation in Obese Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska Lincoln (Other)
Responsible Party: Principal Investigator, Devin Rose, Associate Professor, University of Nebraska Lincoln
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UNebraskaLincolnFDST1
Record Dates: First submitted 2015-11-04; First posted 2015-11-11 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-05

CONDITIONS: Obesity; Overweight
Keywords: Diet; Whole grain; Fruits; Vegetables; Gut health; Anti-inflammatory
MeSH Terms: conditions — Obesity; Overweight | interventions — Fruit; Vegetables; Whole Grains

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Experimental): 3 servings of refined grains per day.
  Interventions: Other: Control
- Fruits and Vegetables (Experimental): 5 servings of fruits and vegetable per day.
  Interventions: Other: Fruits and Vegetables
- Whole Grain (Experimental): 3 servings of whole grains per day.
  Interventions: Other: Whole Grain

INTERVENTIONS:
Other: Fruits and Vegetables — 5 servings of fruits or vegetables
  Arms: Fruits and Vegetables
Other: Whole Grain — 3 servings of whole grain
  Arms: Whole Grain
Other: Control — 3 servings of refined grain
  Arms: Control

SUMMARY:
This study evaluates the impact of increased intake of fruits and vegetables and whole grains on markers of inflammation and gut microbial composition. The treatment groups are 3 servings of whole grain per day; 5 servings of fruits and vegetables per day; and a control (3 servings of refined grains per day provided).

DETAILED DESCRIPTION:
Literature data suggests that fruits and vegetables and whole grains containing dietary fiber and other nutrients are important for maintaining beneficial microbes in the gut. The presence of beneficial microbes in the gut may mediate the subclinical inflammation experienced in metabolic disease. In this project, overweight or obese participants with low intakes of fruits and vegetables or whole grains will increase their intake of these foods to recommended levels. Changes in markers of inflammation and gut microbiota composition will be determined to assess and compare the potential impact of these foods on metabolic disease.

ELIGIBILITY:
Inclusion Criteria:

* Obese or overweight men or women (body mass index, BMI, ≥25 kg/m2)
* Free of known gastrointestinal disease
* No supplements use (excluding multivitamin)
* Participate in less than 1 h of exercise per week
* Have not taken antibiotics in the last six months

Exclusion Criteria:

* Men and women with fruits and vegetable intake exceeding 2 servings/day
* Men and women with whole grain intakes exceeding 1 serving/day
* Pregnant
* Do not fit the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Devin J Rose, PhD, Principal Investigator — University of Nebraska
Locations (1):
- Food Innovation Center, Lincoln, Nebraska, United States

REFERENCES:
- [Derived] Kopf JC, Suhr MJ, Clarke J, Eyun SI, Riethoven JM, Ramer-Tait AE, Rose DJ. Role of whole grains versus fruits and vegetables in reducing subclinical inflammation and promoting gastrointestinal health in individuals affected by overweight and obesity: a randomized controlled trial. Nutr J. 2018 Jul 30;17(1):72. doi: 10.1186/s12937-018-0381-7. PMID 30060746

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Fruits and Vegetables | Whole Grain
Started | 15 | 20 | 17
Completed | 14 | 18 | 17
Not Completed | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Fruits and Vegetables | Whole Grain | Total
Number analyzed (Participants) | 15 | 20 | 17 | 52
Age, Categorical [Count of Participants; unit: Participants] — Population: Only subjects that finished the study were included in the overall analysis.
  Participants
    number analyzed (Participants) | 14 | 18 | 17 | 49
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 13 | 17 | 17 | 47
    >=65 years | 1 | 1 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Only subjects that finished the study were included in the analysis
  years
    number analyzed (Participants) | 14 | 18 | 17 | 49
    (all) | 27.6 (5.9) | 29.4 (12.8) | 39.2 (13.5) | 32.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only subjects that finished the study were included in the analysis
  Participants
    number analyzed (Participants) | 14 | 18 | 17 | 49
    Female | 7 | 12 | 11 | 30
    Male | 7 | 6 | 6 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Interleukin-6 [Mean (Standard Deviation); unit: pg/mL] — Population: Only subjects that finished the study were included in the analysis
  pg/mL
    number analyzed (Participants) | 14 | 18 | 17 | 49
    (all) | 3.6 (2) | 3.8 (2.2) | 4.7 (3.3) | 4.05 (2.58)
high sensitivity C-reactive protein [Mean (Standard Deviation); unit: mg/mL] — Population: Only subjects that finished the study were included in the analysis
  mg/mL
    number analyzed (Participants) | 14 | 18 | 17 | 49
    (all) | 0.65 (0.4) | 0.69 (0.39) | 0.79 (0.56) | 0.71 (0.45)
TNF-alpha [Mean (Standard Deviation); unit: pg/mL] — Population: Only subjects that finished the study were included in the analysis
  pg/mL
    number analyzed (Participants) | 14 | 18 | 17 | 49
    (all) | 23.8 (5.9) | 24.2 (5.2) | 26.7 (4.17) | 24.8 (5.2)
lipopolysaccharide binding protein [Mean (Standard Deviation); unit: mg/L] — Population: Only subjects that finished the study were included in the analysis
  mg/L
    number analyzed (Participants) | 14 | 18 | 17 | 49
    (all) | 1.83 (0.27) | 1.77 (0.45) | 1.90 (0.38) | 1.83 (0.38)

OUTCOME MEASURES:

1. Primary Outcome: Change in Interleukin-6 (Value at Week 8 Minus Value at Week 0)
Description: Plasma samples collected from participants at the beginning (week 0) and end of the study (week 8) will be analyzed for interleukin-6 concentrations using an enzyme linked immunosorbent assay. Changes in the concentrations of these inflammatory markers will be determined from week 0 to week 8.
Time Frame: 8 weeks
Population: IL-6 was analyzed using an ELISA kit. The mean outcome is the mean of difference between the end and beginning of the treatment period.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Control | Fruits and Vegetables | Whole Grain
Number analyzed (Participants) | 14 | 18 | 17
pg/mL | 0.35 (0.45) | -1.08 (0.52) | 0.51 (0.86)
Statistical Analysis 1: Comparison: Control; Test type: Equivalence — Value at week 8 minus value at week 0; p = 0.9942, ANOVA — Corrected for baseline concentrations, age, gender, and body mass index
Statistical Analysis 2: Comparison: Fruits and Vegetables; Test type: Equivalence — Value at week 8 minus value at week 0; p = 0.0062, ANOVA; Corrected for baseline concentrations, age, gender, and body mass index
Statistical Analysis 3: Comparison: Whole Grain; Test type: Equivalence — Value at week 8 minus value at week 0; p = 0.6843, ANOVA; Corrected for baseline concentrations, age, gender, and body mass index

2. Primary Outcome: Change in Tumor Necrosis Factor-α (Value at Week 8 Minus Value at Week 0)
Description: Plasma samples collected from participants at the beginning (week 0) and end of the study (week 8) will be analyzed for tumor necrosis factor-α concentrations using an enzyme linked immunosorbent assay. Changes in the concentrations of these inflammatory markers will be determined from week 0 to week 8.
Time Frame: 8 weeks
Population: TNF-α was analyzed using an ELISA kit. The mean outcome is the mean of difference between the end and beginning of the treatment period.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Control | Fruits and Vegetables | Whole Grain
Number analyzed (Participants) | 14 | 18 | 17
pg/mL | -0.36 (1.58) | -1.11 (1.13) | -5.40 (0.92)
Statistical Analysis 1: Comparison: Control; Test type: Equivalence — Value at week 8 minus value at week 0; p = 0.5096, ANOVA — Corrected for baseline concentrations, age, gender, and body mass index
Statistical Analysis 2: Comparison: Fruits and Vegetables; Test type: Equivalence — Value at week 8 minus value at week 0; p = 0.2276, ANOVA; Corrected for baseline concentrations, age, gender, and body mass index
Statistical Analysis 3: Comparison: Whole Grain; Test type: Equivalence — Value at week 8 minus value at week 0; p = 0.0006, ANOVA; Corrected for baseline concentrations, age, gender, and body mass index

3. Primary Outcome: Change in High Sensitivity C-reactive Protein (Value at Week 8 Minus Value at Week 0)
Description: Plasma samples collected from participants at the beginning (week 0) and end of the study (week 8) will be analyzed for high sensitivity C-reactive protein concentrations using an enzyme linked immunosorbent assay. Changes in the concentrations of these inflammatory markers will be determined from week 0 to week 8.
Time Frame: 8 weeks
Population: C-reactive protein was analyzed using an ELISA kit. The mean outcome is the mean of difference between the end and beginning of the treatment period.
Measure: Mean (Standard Error); unit: mg/mL
Arm/Group | Control | Fruits and Vegetables | Whole Grain
Number analyzed (Participants) | 14 | 18 | 17
mg/mL | 0.01 (0.08) | -0.06 (0.06) | 0.00 (0.12)
Statistical Analysis 1: Comparison: Control; Test type: Equivalence — Value at week 8 minus value at week 0; p = 0.9708, ANOVA — Corrected for baseline concentrations, age, gender, and body mass index
Statistical Analysis 2: Comparison: Fruits and Vegetables; Test type: Equivalence — Value at week 8 minus value at week 0; p = 0.1642, ANOVA; Corrected for baseline concentrations, age, gender, and body mass index
Statistical Analysis 3: Comparison: Whole Grain; Test type: Equivalence — Value at week 8 minus value at week 0; p = 0.6043, ANOVA; Corrected for baseline concentrations, age, gender, and body mass index

4. Primary Outcome: Change in Lipopolysaccharide Binding Protein (Value at Week 8 Minus Value at Week 0)
Description: Plasma samples collected from participants at the beginning (week 0) and end of the study (week 8) will be analyzed for lipopolysaccharide binding protein concentrations using an enzyme linked immunosorbent assay. Changes in the concentrations of these inflammatory markers will be determined from week 0 to week 8.
Time Frame: 8 weeks
Population: Lipopolysaccharide binding protein was analyzed using an ELISA kit. The mean outcome is the mean of difference between the end and beginning of the treatment period.
Measure: Mean (Standard Error); unit: mcg/mL
Arm/Group | Control | Fruits and Vegetables | Whole Grain
Number analyzed (Participants) | 14 | 18 | 17
mcg/mL | 0.14 (0.07) | -0.21 (0.07) | -0.21 (0.08)
Statistical Analysis 1: Comparison: Control; Test type: Equivalence — Value at week 8 minus value at week 0; p = 0.0868, ANOVA — Corrected for baseline concentrations, age, gender, and body mass index
Statistical Analysis 2: Comparison: Fruits and Vegetables; Test type: Equivalence — Value at week 8 minus value at week 0; p = 0.0083, ANOVA; Corrected for baseline concentrations, age, gender, and body mass index
Statistical Analysis 3: Comparison: Whole Grain; Test type: Equivalence — Value at week 8 minus value at week 0; p = 0.0151, ANOVA; Corrected for baseline concentrations, age, gender, and body mass index

5. Secondary Outcome: Change in Gut Microbiota Shannon's Alpha Diversity (Value at Week 8 Minus Value at Week 0)
Description: The Shannon Diversity Index is a quantitative measure that reflects how many different bacterial species there are in a sample. The greater the index, the more diverse the gut microbiota. A negative change indicates a decrease in diversity and a positive change indicates an increase in diversity.
Time Frame: 8 weeks
Population: Alpha diversity was analyzed through the Shannon's Index. The mean outcome is the mean difference between the end and beginning of the treatment period.
Measure: Mean (Standard Error); unit: Shannon's Index
Arm/Group | Control | Fruits and Vegetables | Whole Grain
Number analyzed (Participants) | 14 | 18 | 17
Shannon's Index | 0.05 (0.15) | 0.12 (0.09) | -0.15 (0.12)
Statistical Analysis 1: Comparison: Control; Test type: Equivalence — Value at week 8 minus value at week 0; p = 0.9255, ANOVA — Corrected for baseline concentrations, age, gender, and body mass index
Statistical Analysis 2: Comparison: Fruits and Vegetables; Test type: Equivalence — Value at week 8 minus value at week 0; p = 0.0454, ANOVA; Corrected for baseline concentrations, age, gender, and body mass index
Statistical Analysis 3: Comparison: Whole Grain; Test type: Equivalence — Value at week 8 minus value at week 0; p = 0.2920, ANOVA; Corrected for baseline concentrations, age, gender, and body mass index

6. Secondary Outcome: Change in Fecal Short Chain Fatty Acids (Value at Week 8 Minus Value at Week 0)
Description: Short-chain fatty acids (SCFAs) are the end products of fermentation of dietary fibers by the anaerobic intestinal microbiota. SCFAs have been shown to exert multiple beneficial effects on mammalian energy metabolism.
Time Frame: 8 weeks
Population: Mean outcome is the mean difference between the beginning and end of the study. SCFAs were extracted from stool samples and measured using gas chromatography.
Measure: Mean (Standard Error); unit: mmol/g
Arm/Group | Control | Fruits and Vegetables | Whole Grain
Number analyzed (Participants) | 14 | 18 | 17
mmol/g | -45.82 (22.50) | 10.72 (13.50) | 2.88 (10.18)
Statistical Analysis 1: Comparison: Control; Test type: Equivalence — Value at week 8 minus value at week 0; p = 0.2252, ANOVA — Corrected for baseline concentrations, age, gender, and body mass index
Statistical Analysis 2: Comparison: Fruits and Vegetables; Test type: Equivalence — Value at week 8 minus value at week 0; p = 0.4715, ANOVA; Corrected for baseline concentrations, age, gender, and body mass index
Statistical Analysis 3: Comparison: Whole Grain; Test type: Equivalence — Value at week 8 minus value at week 0; p = 0.7157, ANOVA; Corrected for baseline concentrations, age, gender, and body mass index

7. Secondary Outcome: Change in Branched Chain Fatty Acids (Value at Week 8 Minus Value at Week 0)
Description: Branched chain fatty acids (BCFA) are mostly saturated fatty acids (SFA) with one or more methyl branches on the carbon chain. BCFAs were extracted from stool samples and measured using gas chromatography.
Time Frame: 8 weeks
Population: The outcome mean is the mean difference between the beginning and the end of the study.
Measure: Mean (Standard Error); unit: mmol/g
Arm/Group | Control | Fruits and Vegetables | Whole Grain
Number analyzed (Participants) | 14 | 18 | 17
mmol/g | -0.20 (0.60) | -2.41 (2.79) | 0.16 (0.40)
Statistical Analysis 1: Comparison: Control; Test type: Equivalence — Value at week 8 minus value at week 0; p = 0.8323, ANOVA — Corrected for baseline concentrations, age, gender, and body mass index
Statistical Analysis 2: Comparison: Fruits and Vegetables; Test type: Equivalence — Value at week 8 minus value at week 0; p = 0.8927, ANOVA; Corrected for baseline concentrations, age, gender, and body mass index
Statistical Analysis 3: Comparison: Whole Grain; Test type: Equivalence — Value at week 8 minus value at week 0; p = 0.3173, ANOVA; Corrected for baseline concentrations, age, gender, and body mass index

8. Other Pre Specified Outcome: Change in Body Mass Index (Value at Week 8 Minus Value at Week 0)
Description: Body mass index will be measured on participants at the beginning (week 0) and end of the study (week 8). Changes in body mass index will be determined.
Time Frame: 8 weeks
Population: Weight and height were measured to calculate the BMI. The outcome mean is the mean difference between the beginning and end of the treatment period.
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | Control | Fruits and Vegetables | Whole Grain
Number analyzed (Participants) | 14 | 18 | 17
kg/m^2 | -0.16 (0.09) | -0.22 (0.25) | -0.12 (0.10)
Statistical Analysis 1: Comparison: Control vs Fruits and Vegetables vs Whole Grain; Test type: Equivalence — Value at week 8 minus value at week 0; p = 0.27, ANOVA — Corrected for baseline concentrations, age and gender

ADVERSE EVENTS:
Time Frame: 8 Weeks
Arm/Group | Control | Fruits and Vegetables | Whole Grain
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 0/14 | 0/18 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Statistical Analysis Plan (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/96/NCT02602496/SAP_001.pdf
  • Informed Consent Form (2015-11-05): https://cdn.clinicaltrials.gov/large-docs/96/NCT02602496/ICF_002.pdf
  • Study Protocol (2014-12-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT02602496/Prot_003.pdf